CLINICAL TRIAL: NCT03944200
Title: Randomized, Open Label, Single Oral Administration at Fed State, 2 x 2 Crossover Study to Investigate the Bioequivalence Test of DA-1229_01(A)
Brief Title: A Study to Investigate the Bioequivalence Test of DA-1229_01(A) at Fed State
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dong-A ST Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: DDS18-034BE
Record Dates: First submitted 2019-04-01; First posted 2019-05-09 (Actual); Last update posted 2020-05-20 (Actual); Status verified 2019-05

CONDITIONS: Type2 Diabetes
MeSH Terms: interventions — Drug Evaluation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test drug, Reference drug group (Experimental): Period 1: Single oral administration of 1 tablet of test drug(DA-1229_01(A)) together with 150 mL of water containing 30 g sugar.
  The wash-out for fed study is 7 days. Period 2: Single oral administration of 1 tablet of reference drug(Sugamet SR Tab 5/1000mg®) together with 150 mL of water containing 30 g sugar.
  Interventions: Drug: DA-1229_01(A), Sugamet SR Tab 5/1000mg®
- Reference drug,Test drug group (Active Comparator): Period 1: Single oral administration of 1 tablet of reference drug(Sugamet SR Tab 5/1000mg®) together with 150 mL of water containing 30 g sugar.
  The wash-out for fed study is 7 days. Period 2: Single oral administration of 1 tablet of test drug(DA-1229_01(A)) together with 150 mL of water containing 30 g sugar.
  Interventions: Drug: Sugamet SR Tab 5/1000mg®, DA-1229_01(A)

INTERVENTIONS:
Drug: DA-1229_01(A), Sugamet SR Tab 5/1000mg® — Period 1: Single oral administration of 1 tablet of test drug(DA-1229_01(A)) together with 150 mL of water containing 30 g sugar.
  The wash-out for fed study is 7 days. Period 2: Single oral administration of 1 tablet of reference drug(Sugamet SR Tab 5/1000mg®) together with 150 mL of water containing 30 g sugar.
  Other Names: Test drug, Reference drug group
  Arms: Test drug, Reference drug group
Drug: Sugamet SR Tab 5/1000mg®, DA-1229_01(A) — Period 1: Single oral administration of 1 tablet of reference drug(Sugamet SR Tab 5/1000mg®) together with 150 mL of water containing 30 g sugar.
  The wash-out for fed study is 7 days. Period 2: Single oral administration of 1 tablet of test drug(DA-1229_01(A)) together with 150 mL of water containing 30 g sugar.
  Other Names: Reference drug,Test drug group
  Arms: Reference drug,Test drug group

SUMMARY:
A study demonstrates the bioequivalence of DA-1229_01(A) at Fed State when compared with Sugamet sustained-release(SR) Tab 5/1000mg® in healthy adults

ELIGIBILITY:
Inclusion Criteria:

* Adult patients over 19 years of age at the time of health examination
* Female patients who were confirmed to be not pregnant at health examination
* Patients without a history of mental illness in the past 5 years

Exclusion Criteria:

* Patients who have taken medications which could affect the results of the clinical trial in the past 10 days of participating in the clinical trial
* Patients with a congestive heart failure which requires medicinal treatment
* Patients who have made a whole blood donation in the past 2 months or an apheresis donation in the past 2 weeks of participating in the clinical trial
* Female patients who are lactating

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-02-07 (Actual); Primary Completion 2019-03-25 (Actual); Study Completion 2019-03-25 (Actual)

PRIMARY OUTCOMES:
Area under the concentration-time curve(AUCt) | Hour -1 ~ Hour 24
  AUCt of metformin
Maximum plasmaconcentration of drug in plasma(Cmax) | Hour -1 ~ Hour 24
  Cmax of metformin

SECONDARY OUTCOMES:
Area under the plasma drug concentration-time curve from time 0 to infinity(AUCinf) | Hour -1 ~ Hour 24
  AUCinf of metformin
AUCt/AUCinf | Hour -1 ~ Hour 24
  AUCt/AUCinf of metformin
Time to reach the maximum plasma concentration(Tmax) | Hour -1 ~ Hour 24
  Tmax of metformin
Terminal elimination rate constant(ramda z) | Hour -1 ~ Hour 24
  ramda z of metformin
Terminal elimination half-life(t1/2) | Hour -1 ~ Hour 24
  t1/2 of metformin

CONTACTS AND LOCATIONS:
Overall Officials: Sung Dae Kwon, M.D., Ph.D., Principal Investigator — Metro Hospital
Locations (1):
- Metro Hospital, Anyang-si, Gyeonggi-do, South Korea